CLINICAL TRIAL: NCT04991727
Title: Pulmonary Ultrasound to Evaluate Protective Lung Ventilation in Obese Patients With Postoperative Pulmonary Complications Impact
Brief Title: Evaluation of Protective Pulmonary Ventilation by Pulmonary Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-2021-277
Record Dates: First submitted 2021-06-26; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Assessment
Keywords: lung ultrasound; Protective pulmonary ventilation; Postoperative pulmonary complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEEP: The patient was admitted to the operating room, and routine ECG monitoring was performed. The patient was placed in supine position, and ultrasound lung examination was performed. The images of the patient were saved and the score of lung ventilation area was recorded. The induction of general anesthesia was started, and endotracheal intubation was performed after 3min of preoxygenation (100% O2) to establish a safe and effective artificial airway.Mechanical ventilation was performed after endotracheal intubation, and a second time was performed immediately after endotracheal intubation was completed.Pulmonary ultrasound was performed. The PEEPgroup was given the first RM (pulmonary retraction) with pressure maintained at 40cmH2O for 30s, followed by a 7cmH2O PEEP to maintain mechanical ventilation, and the RMS was repeated every 30 minutes until the end of surgery
  Interventions: Behavioral: recruitment maneuvers
- ZEEP: The patient was admitted to the operating room, and routine ECG monitoring was performed. The patient was placed in supine position, and ultrasound lung examination was performed. The images of the patient were saved and the score of lung ventilation area was recorded. The induction of general anesthesia was started, and endotracheal intubation was performed after 3min of preoxygenation (100% O2) to establish a safe and effective artificial airway. Mechanical ventilation was performed after endotracheal intubation, and a second time was performed immediately after endotracheal intubation was completed
  On pulmonary ultrasound, patients in the ZEEP group maintained normal mechanical ventilation throughout the operation without PEEP or RMS
  Interventions: Behavioral: recruitment maneuvers

INTERVENTIONS:
Behavioral: recruitment maneuvers — Immediately after endotracheal intubation is completed
  First RM (pulmonary retraction), maintain pressure at 40cmH2O for 30s, and then
  Mechanical ventilation was maintained with 7cmH2O PEEP, and the RMS was repeated every 30 minutes until the end of surgery

SUMMARY:
Peri - operative ultrasonography was used to evaluate the effects of protective lung ventilation on the postoperative lungs of obese patients.The purpose of this study was to apply ultrasound lung ventilation area score to the monitoring of pulmonary complications in patients with postoperative obesity.To verify the reliability and practicability of perioperative lung ultrasound quantitative scoring.

DETAILED DESCRIPTION:
Ultrasound lung ventilation area score was applied to monitor the pulmonary complications of patients after obesity operation to verify the perioperative period.

The reliability and practicability of quantitative lung ultrasound score to clarify the effect of protective lung ventilation under perioperative pulmonary ultrasound monitoring on obesity patients.To guide the management of mechanical ventilation under general anesthesia and the prevention and treatment of postoperative pulmonary complications

ELIGIBILITY:
Inclusion Criteria:

* enrollment of patients aged 18 years or above；
* Eligible adult patients had an American Society of Anesthesiologists (ASA) physical status classification of I to IV
* undergoing elective or expedited nonurgent, noncardiac surgery with general anesthesia

Exclusion Criteria:

* patient refusal;
* morbid obesity (BMI >40 kg/ m²);
* American Society of Anesthesiologists (ASA) physical status categories IV-V;
* previous intrathoracic procedure;
* severechronic obstructive pulmonary disease (forced expiratory volume in 1 s <30% of the predicted value;
* a contraindication to radial artery cannulation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery, non-cardiac surgery, in the Heart and Brain Hospital of Ningxia Medical University from June, 2021 to October, 2023
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-21 (Estimated); Primary Completion 2023-10-23 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Lung ultrasound scoring | in the morning of the first day
  Four signs were used in lung ultrasound scoring
  Lung ultrasound score: N (0): pleural line and A line, less than 3 B lines; B1 (1 mark): More than 3
  B line; B2 (2 points): Fuse line B; C (3 points): Signs of lung consolidation. The higher the score is, the worse the pulmonary ventilation status is.
  When scoring, the sign with the greatest severity is taken as the score value of the examination area. There are 12 examination areas in both lungs, so we have a LUS
  The score is between 0 and 36

SECONDARY OUTCOMES:
Results of arterial blood gas analysis | entering the operating room, in the morning of the first day ,the second day , the third day after surgery
  PCO2
Mechanical ventilation parameter | entering the operating room, in the morning of the first day ,the second day , the third day after surgery
  peak inspiratory pressure

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

REFERENCES:
- [Background] Wanguemert Perez AL. Clinical applications of pulmonary ultrasound. Med Clin (Barc). 2020 Apr 10;154(7):260-268. doi: 10.1016/j.medcli.2019.11.001. Epub 2020 Jan 8. English, Spanish. PMID 31926654
- [Background] Costamagna A, Pivetta E, Goffi A, Steinberg I, Arina P, Mazzeo AT, Del Sorbo L, Veglia S, Davini O, Brazzi L, Ranieri VM, Fanelli V. Clinical performance of lung ultrasound in predicting ARDS morphology. Ann Intensive Care. 2021 Mar 29;11(1):51. doi: 10.1186/s13613-021-00837-1. PMID 33779834